CLINICAL TRIAL: NCT00467389
Title: Donepezil Effects on Cocaine Craving and Pharmacokinetics
Brief Title: Use of Donepezil for Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEUA-014-05S
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Cocaine Abuse and Dependence
Keywords: Acetylcholine; Acetylcholinesterase; Butyrylcholinesterase; Cholinesterase Inhibitor
MeSH Terms: conditions — Cocaine-Related Disorders; Pain; Butyrylcholinesterase deficiency | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Placebo First (Experimental): Three days of daily treatment with oral placebo, followed by three days of daily treatment with 5 mg of donepezil
  Interventions: Drug: Donepezil, 5 mg daily; Other: Oral Placebo
- Donepezil First (Experimental): Three days of daily treatment with 5 mg of donepezil, followed by three days of daily treatment with oral placebo.
  Interventions: Drug: Donepezil, 5 mg daily; Other: Oral Placebo

INTERVENTIONS:
Drug: Donepezil, 5 mg daily — This is a commercially available cholinesterase inhibitor that is approved for use in Alzheimer's disease.
  Other Names: Aricept
Other: Oral Placebo — Inactive Comparator with Similar Appearance to Active Medication
  Other Names: Inactive Comparator

SUMMARY:
The purpose of this study is to determine the safety of intravenous cocaine in subjects receiving oral donepezil.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, placebo controlled, inpatient, single-center, parallel group evaluation of the potential for oral donepezil to attenuate cocaine-induced craving. Non-treatment-seeking cocaine-experienced volunteers will receive baseline treatment with intravenous cocaine (30Mg). Forty-two subjects that tolerate baseline cocaine infusions will then receive two subsequent intravenous doses of cocaine during double-blind treatment with oral placebo or 5 mg daily of donepezil. Each dose of cocaine will be preceded or followed by administration of intravenous placebo (saline) in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Non-treatment seeking, experienced cocaine users, who have used cocaine by smoking or intravenous injection within the four weeks prior to screening, and must supply a cocaine-positive urine obtained within four weeks of entry into the study.

Exclusion Criteria:

* Shows signs of psychostimulant toxicity, or has a history of a medical adverse reaction to cocaine or other psychostimulants, including loss of consciousness, chest pain, cardiac ischemia, or seizure.
* Has a current psychiatric disorder other than drug abuse or dependence or dementia.
* Meets the Diagnostic and Statistical Manual of Mental Disorders-IV criteria for dependence to opiates, benzodiazepines, alcohol, or other sedative-hypnotics.
* Has received opiate-substitution therapy (methadone or buprenorphine) within two months prior to enrollment.
* Has current or past history of seizure disorder, including alcohol- or psychostimulant- related seizures, or family history of seizure disorder.
* Has a diagnosis of adult asthma, or chronic obstructive pulmonary disease, including a history of acute asthma within the past two years, and those with current or recent (with the past two years) treatment with an inhaled or oral beta-adrenergic agonist.
* Has had head trauma that resulted in neurological sequelae.
* Has an unstable medical condition, which, in the judgement of investigators, would make participation hazardous.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Grasing, MD, Principal Investigator — VA Medical Center
Locations (1):
- VA Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Result] Grasing K, Mathur D, Newton TF, DeSouza C. Donepezil treatment and the subjective effects of intravenous cocaine in dependent individuals. Drug Alcohol Depend. 2010 Feb 1;107(1):69-75. doi: 10.1016/j.drugalcdep.2009.09.010. PMID 19836169

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Treatment First: Participants initially treated with oral placebo, and later treated with oral donepezil
- Donepezil Treatment First: Participants initially treated with oral donepezil, and later treated with oral placebo
Period: Overall Study
Arm/Group | Placebo Treatment First | Donepezil Treatment First
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participating subjects
Groups:
- All Participants: All recruited subjects
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.4 (0.8)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Safety in Subjects Receiving Donepezil
Description: Patients evaluated for clinical and laboratory adverse events
Time Frame: Two weeks
Population: All participants included
Measure: Number; unit: Participants with an Adverse Event
Groups:
- Placebo Treatment Period: Inactive Comparator
- Donepezil Treatment Period: Active Treatment
Arm/Group | Placebo Treatment Period | Donepezil Treatment Period
Number analyzed (Participants) | 12 | 12
Participants with an Adverse Event | 0 | 2

2. Secondary Outcome: Cocaine Subjective Effects
Description: Cocaine Induced 'High' by VAS (visual analogue scale, between 3 and 30 minutes after intravenous dosing, in mm). VAS results ranged from 0 (minimum effect) to 100 (maximum effect).
Time Frame: 3 to 30 minutes
Measure: Mean (Standard Error); unit: mm
Arm/Group | Placebo Treatment Period | Donepezil Treatment Period
Number analyzed (Participants) | 12 | 12
mm | 44.1 (17.8) | 89.9 (35.3)

3. Secondary Outcome: Cocaine Pharmacokinetics
Description: Area-Under-the-Curve for Plasma Concentration
Time Frame: 0 to 8 hours
Measure: Mean (Standard Error); unit: ng-hr/ml
Arm/Group | Placebo Treatment Period | Donepezil Treatment Period
Number analyzed (Participants) | 12 | 12
ng-hr/ml | 34,503 (3,599) | 40,812 (5,244)

ADVERSE EVENTS:
Arm/Group | Placebo Treatment Period | Donepezil Treatment Period
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Period (N=12) | Donepezil Treatment Period (N=12)
Gastrointestinal distress (Gastrointestinal disorders) | 0 (0) | 1 (1) — One patient experienced a single episode of nausea and vomiting on his second day of treatment with donepezil that resolved spontaneously.
Chest discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) — An additional patient reported 5 minutes of mild chest discomfort that he attributed to eating too much during his third day of donepezil treatment, with no electrocardiogram changes observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes